CLINICAL TRIAL: NCT05392205
Title: Evaluating the Potential Usefulness of 68Ga-FAP-2286 PET/CT in Patients With Various Types of Cancer and Compared With 18F-FDG PET/CT
Brief Title: Comaprison of 68Ga-FAP-2286 and 18F-FDG PET/CT in Patients With Various Types of Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022KY013
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2022-03

CONDITIONS: Tumor, Solid; Positron-Emission Tomography
Keywords: Tumor; Solid; Positron-Emission Tomography; diagnosis
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAP-2286 (Experimental): Each subject receives a single intravenous injection of 18F-FDG and 68Ga-FAP-2286, and undergo PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: 18F-FDG

INTERVENTIONS:
Diagnostic Test: 18F-FDG — Each subject receives a single intravenous injection of 18F-FDG and 68Ga-FAP-2286, and undergo PET/CT imaging within the specified time. A part of participants will also undergo additional 68Ga-FAPI-46 PET/CT for comparison.

SUMMARY:
To evaluate the potential usefulness of 68Ga-FAP-2286 positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various types of cancer, and compared with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Subjects with various types of cancer underwent contemporaneous 68Ga-FAP-2286 and 18F-FDG PET/CT either for an initial assessment or for recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The numbers of positive tumor lesions of 18F-FDG and 68Ga-FAP-2286 PET/CT were recorded by visual interpretation. The sensitivity, specificity, and accuracy of 68Ga-FAP-2286, 18F-FDG PET/CT were calculated and compared to evaluate the diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 years or order);
* patients with suspected or newly diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report);
* patients who had scheduled both 18F-FDG and 68Ga-FAP-2286 PET/CT scans;
* patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* patients with non-malignant lesions;
* patients with pregnancy;
* the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 90 days
  The sensitivity, specificity, and accuracy of 18F-FDG and 68Ga-FAP-2286 PET/CT were calculated and compared to evaluate the diagnostic efficacy.

SECONDARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of 18F-FDG and 68Ga-FAP-2286 PET/CT for each target lesion of subject or suspected primary tumor or/and metastasis.
Number of lesions | 90 days
  The numbers of positive primary and metastatic lesions of 18F-FDG and 68Ga-FAP-2286 PET/CT were recorded by visual interpretation.

CONTACTS AND LOCATIONS:
Overall Officials: Long Sun, PhD, Study Director — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First affiliated hospital of xiamen university, Xiamen, Fujian, China